CLINICAL TRIAL: NCT05224596
Title: Gastric Cancer Detection by Liquid Biopsy in Peripheral Blood: A Prospective Study
Brief Title: AssesSment of Early-deteCtion basEd oN liquiD Biopsy in GASTRIC Cancer, ASCEND-Gastric
Acronym: ASCEND-Gastric
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Guangzhou Burning Rock Bioengineering Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: B2020-390R
Record Dates: First submitted 2022-01-05; First posted 2022-02-04 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Cancer
Keywords: Cancer; liquid biopsy; cell-free DNA (cfDNA) methylation; circulating tumor DNA (ctDNA) mutation; whole blood miRNA
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Baseline blood samples will be collected from new diagnosis cancer participants.
  Interventions: Diagnostic Test: Blood draw and blood-based biomarkers analyses
- Benign disease arm: Baseline blood samples will be collected from new diagnosis benign gastric disease participants.
  Interventions: Diagnostic Test: Blood draw and blood-based biomarkers analyses

INTERVENTIONS:
Diagnostic Test: Blood draw and blood-based biomarkers analyses — blood-based biomarkers analyses

SUMMARY:
ASCEND-Gastric is a prospective, multi-omics, observational study aimed at detecting gastric cancer by combined assays for serum protein markers, deep sequencing of cell-free DNA (cfDNA), circulating tumor DNA (ctDNA) mutation and circulating RNA. The study will enroll 498 participants, including 128 patients with benign gastric diseases and 370 patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Age 40-75 years at the day of consenting to the study.
* Able to provide a written informed consent.
* No prior cancer treatment (local or systematic) with either of the following:

A. Pathologically confirmed cancer diagnosis within 42 days prior to blood draw.

B. High suspicious for cancer diagnosis by imaging tests or other routine clinical examinations, with confirmed pathological cancer diagnosis within 42 days after the blood draw.

Exclusion Criteria for Cancer Arm Participants:

* Insufficient qualified blood samples.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 7 days prior to blood draw.
* Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw.
* With other known malignant tumors or multiple primary tumors.

Inclusion Criteria for Benign Disease Arm Participants:

* Age 40-75 years at the day of consenting to the study.
* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* Have either of the following:

A. Pathological confirmed diagnosis of benign diseases within 90 days prior to the study blood draw, with no prior treatment such as surgical resection.

B. High suspicious for benign diseases diagnosis by radiological or other routine clinical assessments, with confirmed benign diseases diagnosis within 42 days after study blood draw.

Exclusion Criteria for Benign Disease Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 7 days prior to study blood draw.
* Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants in cancer arm will be recruited with new diagnosis of gastric cancer and without any types of tumor treatment.
  Eligible participants in benign disease arm will be recruited with new diagnosis of benign gastric disease and without any types of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-09-22 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the cfDNA methylation-based model in detecting gastric cancer. | 30 months

SECONDARY OUTCOMES:
The differences of sensitivity and specificity in gastric cancer participants at different clinical stages. | 30 months
Sensitivity and specificity for detecting gastric cancer of a cfDNA methylation-based model, in combination with other biomarkers. | 30 months
Sensitivity and specificity of a ctDNA mutation-based model and a serum protein-based model in detecting gastric cancer, respectively. | 30 months

OTHER OUTCOMES:
Sensitivity and specificity of a blood miRNA-based model in detecting gastric cancer. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Sun Sun, MD, Principal Investigator — Zhongshan Hospital, Fudan University,China; Xuefei Wang, MD, Principal Investigator — Zhongshan Hospital, Fudan University,China
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Sano T, Coit DG, Kim HH, Roviello F, Kassab P, Wittekind C, Yamamoto Y, Ohashi Y. Proposal of a new stage grouping of gastric cancer for TNM classification: International Gastric Cancer Association staging project. Gastric Cancer. 2017 Mar;20(2):217-225. doi: 10.1007/s10120-016-0601-9. Epub 2016 Feb 20. PMID 26897166
- [Background] So JBY, Kapoor R, Zhu F, Koh C, Zhou L, Zou R, Tang YC, Goo PCK, Rha SY, Chung HC, Yoong J, Yap CT, Rao J, Chia CK, Tsao S, Shabbir A, Lee J, Lam KP, Hartman M, Yong WP, Too HP, Yeoh KG. Development and validation of a serum microRNA biomarker panel for detecting gastric cancer in a high-risk population. Gut. 2021 May;70(5):829-837. doi: 10.1136/gutjnl-2020-322065. Epub 2020 Oct 7. PMID 33028667
- [Background] Miki K. Gastric cancer screening using the serum pepsinogen test method. Gastric Cancer. 2006;9(4):245-53. doi: 10.1007/s10120-006-0397-0. Epub 2006 Nov 24. PMID 17235625
- [Background] Li MY, Zhang DQ, Lu X, Chen WC. [Comparison of two serological methods in screening gastric cancer and its precancerous condition]. Zhonghua Nei Ke Za Zhi. 2018 Dec 1;57(12):907-911. doi: 10.3760/cma.j.issn.0578-1426.2018.12.006. Chinese. PMID 30486559
- [Background] Hamashima C; Systematic Review Group and Guideline Development Group for Gastric Cancer Screening Guidelines. Update version of the Japanese Guidelines for Gastric Cancer Screening. Jpn J Clin Oncol. 2018 Jul 1;48(7):673-683. doi: 10.1093/jjco/hyy077. PMID 29889263
- [Background] Choi KS, Jun JK, Park EC, Park S, Jung KW, Han MA, Choi IJ, Lee HY. Performance of different gastric cancer screening methods in Korea: a population-based study. PLoS One. 2012;7(11):e50041. doi: 10.1371/journal.pone.0050041. Epub 2012 Nov 29. PMID 23209638
- [Background] Zhang X, Li M, Chen S, Hu J, Guo Q, Liu R, Zheng H, Jin Z, Yuan Y, Xi Y, Hua B. Endoscopic Screening in Asian Countries Is Associated With Reduced Gastric Cancer Mortality: A Meta-analysis and Systematic Review. Gastroenterology. 2018 Aug;155(2):347-354.e9. doi: 10.1053/j.gastro.2018.04.026. Epub 2018 Apr 30. PMID 29723507
- [Background] Chen M, Zhao H. Next-generation sequencing in liquid biopsy: cancer screening and early detection. Hum Genomics. 2019 Aug 1;13(1):34. doi: 10.1186/s40246-019-0220-8. PMID 31370908
- [Background] Kang HM, Kim GH, Jeon HK, Kim DH, Jeon TY, Park DY, Jeong H, Chun WJ, Kim MH, Park J, Lim M, Kim TH, Cho YK. Circulating tumor cells detected by lab-on-a-disc: Role in early diagnosis of gastric cancer. PLoS One. 2017 Jun 29;12(6):e0180251. doi: 10.1371/journal.pone.0180251. eCollection 2017. PMID 28662130
- [Background] Haber DA, Velculescu VE. Blood-based analyses of cancer: circulating tumor cells and circulating tumor DNA. Cancer Discov. 2014 Jun;4(6):650-61. doi: 10.1158/2159-8290.CD-13-1014. Epub 2014 May 6. PMID 24801577
- [Background] Cristiano S, Leal A, Phallen J, Fiksel J, Adleff V, Bruhm DC, Jensen SO, Medina JE, Hruban C, White JR, Palsgrove DN, Niknafs N, Anagnostou V, Forde P, Naidoo J, Marrone K, Brahmer J, Woodward BD, Husain H, van Rooijen KL, Orntoft MW, Madsen AH, van de Velde CJH, Verheij M, Cats A, Punt CJA, Vink GR, van Grieken NCT, Koopman M, Fijneman RJA, Johansen JS, Nielsen HJ, Meijer GA, Andersen CL, Scharpf RB, Velculescu VE. Genome-wide cell-free DNA fragmentation in patients with cancer. Nature. 2019 Jun;570(7761):385-389. doi: 10.1038/s41586-019-1272-6. Epub 2019 May 29. PMID 31142840
- [Background] Cabel L, Decraene C, Bieche I, Pierga JY, Bennamoun M, Fuks D, Ferraz JM, Lefevre M, Baulande S, Bernard V, Vacher S, Mariani P, Proudhon C, Bidard FC, Louvet C. Limited Sensitivity of Circulating Tumor DNA Detection by Droplet Digital PCR in Non-Metastatic Operable Gastric Cancer Patients. Cancers (Basel). 2019 Mar 21;11(3):396. doi: 10.3390/cancers11030396. PMID 30901876
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Cree IA, Uttley L, Buckley Woods H, Kikuchi H, Reiman A, Harnan S, Whiteman BL, Philips ST, Messenger M, Cox A, Teare D, Sheils O, Shaw J; UK Early Cancer Detection Consortium. The evidence base for circulating tumour DNA blood-based biomarkers for the early detection of cancer: a systematic mapping review. BMC Cancer. 2017 Oct 23;17(1):697. doi: 10.1186/s12885-017-3693-7. PMID 29061138
- [Background] Cohen JD, Javed AA, Thoburn C, Wong F, Tie J, Gibbs P, Schmidt CM, Yip-Schneider MT, Allen PJ, Schattner M, Brand RE, Singhi AD, Petersen GM, Hong SM, Kim SC, Falconi M, Doglioni C, Weiss MJ, Ahuja N, He J, Makary MA, Maitra A, Hanash SM, Dal Molin M, Wang Y, Li L, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Goggins MG, Hruban RH, Wolfgang CL, Klein AP, Tomasetti C, Papadopoulos N, Kinzler KW, Vogelstein B, Lennon AM. Combined circulating tumor DNA and protein biomarker-based liquid biopsy for the earlier detection of pancreatic cancers. Proc Natl Acad Sci U S A. 2017 Sep 19;114(38):10202-10207. doi: 10.1073/pnas.1704961114. Epub 2017 Sep 5. PMID 28874546
- [Background] Cohen JD, Li L, Wang Y, Thoburn C, Afsari B, Danilova L, Douville C, Javed AA, Wong F, Mattox A, Hruban RH, Wolfgang CL, Goggins MG, Dal Molin M, Wang TL, Roden R, Klein AP, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Vogelstein JT, Browne JD, Schoen RE, Brand RE, Tie J, Gibbs P, Wong HL, Mansfield AS, Jen J, Hanash SM, Falconi M, Allen PJ, Zhou S, Bettegowda C, Diaz LA Jr, Tomasetti C, Kinzler KW, Vogelstein B, Lennon AM, Papadopoulos N. Detection and localization of surgically resectable cancers with a multi-analyte blood test. Science. 2018 Feb 23;359(6378):926-930. doi: 10.1126/science.aar3247. Epub 2018 Jan 18. PMID 29348365
- [Background] Klutstein M, Nejman D, Greenfield R, Cedar H. DNA Methylation in Cancer and Aging. Cancer Res. 2016 Jun 15;76(12):3446-50. doi: 10.1158/0008-5472.CAN-15-3278. Epub 2016 Jun 2. PMID 27256564
- [Background] Meng H, Cao Y, Qin J, Song X, Zhang Q, Shi Y, Cao L. DNA methylation, its mediators and genome integrity. Int J Biol Sci. 2015 Apr 8;11(5):604-17. doi: 10.7150/ijbs.11218. eCollection 2015. PMID 25892967
- [Background] Morgan AE, Davies TJ, Mc Auley MT. The role of DNA methylation in ageing and cancer. Proc Nutr Soc. 2018 Nov;77(4):412-422. doi: 10.1017/S0029665118000150. Epub 2018 Apr 30. PMID 29708096
- [Background] Widschwendter M, Jones A, Evans I, Reisel D, Dillner J, Sundstrom K, Steyerberg EW, Vergouwe Y, Wegwarth O, Rebitschek FG, Siebert U, Sroczynski G, de Beaufort ID, Bolt I, Cibula D, Zikan M, Bjorge L, Colombo N, Harbeck N, Dudbridge F, Tasse AM, Knoppers BM, Joly Y, Teschendorff AE, Pashayan N; FORECEE (4C) Consortium. Epigenome-based cancer risk prediction: rationale, opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):292-309. doi: 10.1038/nrclinonc.2018.30. Epub 2018 Feb 27. PMID 29485132
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436
- [Background] Church TR, Wandell M, Lofton-Day C, Mongin SJ, Burger M, Payne SR, Castanos-Velez E, Blumenstein BA, Rosch T, Osborn N, Snover D, Day RW, Ransohoff DF; PRESEPT Clinical Study Steering Committee, Investigators and Study Team. Prospective evaluation of methylated SEPT9 in plasma for detection of asymptomatic colorectal cancer. Gut. 2014 Feb;63(2):317-25. doi: 10.1136/gutjnl-2012-304149. Epub 2013 Feb 13. PMID 23408352
- [Background] Hu W, Zheng W, Liu Q, Chu H, Chen S, Kim JJ, Wu J, Si J. Diagnostic accuracy of DNA methylation in detection of gastric cancer: a meta-analysis. Oncotarget. 2017 Nov 3;8(68):113142-113152. doi: 10.18632/oncotarget.22613. eCollection 2017 Dec 22. PMID 29348893
- [Background] Anderson BW, Suh YS, Choi B, Lee HJ, Yab TC, Taylor WR, Dukek BA, Berger CK, Cao X, Foote PH, Devens ME, Boardman LA, Kisiel JB, Mahoney DW, Slettedahl SW, Allawi HT, Lidgard GP, Smyrk TC, Yang HK, Ahlquist DA. Detection of Gastric Cancer with Novel Methylated DNA Markers: Discovery, Tissue Validation, and Pilot Testing in Plasma. Clin Cancer Res. 2018 Nov 15;24(22):5724-5734. doi: 10.1158/1078-0432.CCR-17-3364. Epub 2018 May 29. PMID 29844130
- [Background] Gao Y, Zhang K, Xi H, Cai A, Wu X, Cui J, Li J, Qiao Z, Wei B, Chen L. Diagnostic and prognostic value of circulating tumor DNA in gastric cancer: a meta-analysis. Oncotarget. 2017 Jan 24;8(4):6330-6340. doi: 10.18632/oncotarget.14064. PMID 28009985
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Chen X, Gole J, Gore A, He Q, Lu M, Min J, Yuan Z, Yang X, Jiang Y, Zhang T, Suo C, Li X, Cheng L, Zhang Z, Niu H, Li Z, Xie Z, Shi H, Zhang X, Fan M, Wang X, Yang Y, Dang J, McConnell C, Zhang J, Wang J, Yu S, Ye W, Gao Y, Zhang K, Liu R, Jin L. Non-invasive early detection of cancer four years before conventional diagnosis using a blood test. Nat Commun. 2020 Jul 21;11(1):3475. doi: 10.1038/s41467-020-17316-z. PMID 32694610